CLINICAL TRIAL: NCT01884805
Title: Feasibility of Measurement of Optical Aberrations in Hyperopia by Using an Adaptive Optics Visual Simulator (AOVIS-I)
Acronym: HyperVOPTICA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Centre de Référence National du Kératocône (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12 483 03
Record Dates: First submitted 2013-05-24; First posted 2013-06-24 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Hyperopia
Keywords: Adaptive Optics Visual Simulator; Wavefront aberrometer; Optical Aberrations; Hyperopia
MeSH Terms: conditions — Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Monocular Adaptive Optics Visual Simulator (AOVIS-I) (Other)
  Interventions: Device: Monocular Adaptive Optics Visual Simulator (AOVIS-I)

INTERVENTIONS:
Device: Monocular Adaptive Optics Visual Simulator (AOVIS-I) — The procedure is guided by the custom made software and its graphical user interface. The interface has been designed to be user-friendly, being very similar to the software usually managed by the clinicians in their daily professional practice. The complete procedure in one patient takes less than 5 minutes and is completely non-invasive. The optical measurements only involve the use of low power infrared laser and the visual testing is as simple for the patients as watching television and making responses.

SUMMARY:
The primary purpose of the protocol is to evaluate the adaptive optics visual simulator to measure optical aberrations in hyperopic eyes.

The study hypotheses are the:

* Ability to measure optical aberrations in hypermetropia.
* Knowledge of optical aberrations of the eye hyperopic.
* To adapt therapeutic management in optical aberrations measured.

DETAILED DESCRIPTION:
The procedure is guided by the custom made software and its graphical user interface. The interface has been designed to be user-friendly, being very similar to the software usually managed by the clinicians in their daily professional practice. The complete procedure in one patient takes less than 5 minutes and is completely non-invasive. The optical measurements only involve the use of low power infrared laser and the visual testing is as simple for the patients as watching television and making responses.

ELIGIBILITY:
Inclusion Criteria:

* hyperopic patients
* to be able to understand an information and give a consent
* affiliated to medical insurance

Exclusion Criteria:

* pregnant women or nursing mothers
* ocular infection
* keratitis
* restless patients
* ocular surgery 90 days before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Measurement of optical aberrations | 1 day (Participants will be followed for the duration of ophtalmology consultation)
  Feasibility of Measurement of optical aberrations in hyperopia by using an Adaptive Optics Visual Simulator AOVIS-I. Outcome measure is assessed during a consultation

SECONDARY OUTCOMES:
Reproductibility of the measures | 1 day (Participants will be followed for the duration of ophtalmology consultation)
  Evaluate the reproducibility of the measures obtained in hyperopic eyes. Outcome measure is assessed during a consultation
Quantitative measurement of optical aberrations | 1 day (Participants will be followed for the duration of ophtalmology consultation)
  Expression of optical aberrations in numerical measures. Outcome measure is assessed during a consultation

CONTACTS AND LOCATIONS:
Overall Officials: François MALECAZE, PHD, Principal Investigator
Locations (1):
- University Hospital, Toulouse, Toulouse, Midi-Pyrenees, France

REFERENCES:
- [Background] Fernandez EJ, Manzanera S, Piers P, Artal P. Adaptive optics visual simulator. J Refract Surg. 2002 Sep-Oct;18(5):S634-8. doi: 10.3928/1081-597X-20020901-27. PMID 12361172
- [Background] Piers PA, Fernandez EJ, Manzanera S, Norrby S, Artal P. Adaptive optics simulation of intraocular lenses with modified spherical aberration. Invest Ophthalmol Vis Sci. 2004 Dec;45(12):4601-10. doi: 10.1167/iovs.04-0234. PMID 15557473
- [Background] Piers PA, Manzanera S, Prieto PM, Gorceix N, Artal P. Use of adaptive optics to determine the optimal ocular spherical aberration. J Cataract Refract Surg. 2007 Oct;33(10):1721-6. doi: 10.1016/j.jcrs.2007.08.001. PMID 17889766
- [Background] Manzanera S, Prieto PM, Ayala DB, Lindacher JM, Artal P. Liquid crystal Adaptive Optics Visual Simulator: Application to testing and design of ophthalmic optical elements. Opt Express. 2007 Nov 26;15(24):16177-88. doi: 10.1364/oe.15.016177. PMID 19550905
- [Background] Villegas EA, Alcon E, Artal P. Optical quality of the eye in subjects with normal and excellent visual acuity. Invest Ophthalmol Vis Sci. 2008 Oct;49(10):4688-96. doi: 10.1167/iovs.08-2316. Epub 2008 Jun 14. PMID 18552387
- [Background] Fernandez EJ, Prieto PM, Artal P. Wave-aberration control with a liquid crystal on silicon (LCOS) spatial phase modulator. Opt Express. 2009 Jun 22;17(13):11013-25. doi: 10.1364/oe.17.011013. PMID 19550501
- [Background] Fernandez EJ, Prieto PM, Artal P. Binocular adaptive optics visual simulator. Opt Lett. 2009 Sep 1;34(17):2628-30. doi: 10.1364/OL.34.002628. PMID 19724513
- [Background] Perez GM, Manzanera S, Artal P. Impact of scattering and spherical aberration in contrast sensitivity. J Vis. 2009 Mar 25;9(3):19.1-10. doi: 10.1167/9.3.19. PMID 19757958
- [Background] Bueno JM, Acosta E, Schwarz C, Artal P. Wavefront measurements of phase plates combining a point-diffraction interferometer and a Hartmann-Shack sensor. Appl Opt. 2010 Jan 20;49(3):450-6. doi: 10.1364/AO.49.000450. PMID 20090810